CLINICAL TRIAL: NCT01645267
Title: Calcaneal Neck Lengthening Osteotomy - Allogen Bone Graft Material Versus a Hydroxyappatite / β- Tricalcium Phosphate Bone Substitute
Brief Title: Calcaneal Neck Lengthening Osteotomy With Artificial Bone Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Martin Gottliebsen, PhD-student, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-20090162
Record Dates: First submitted 2012-07-12; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Flatfoot
MeSH Terms: conditions — Flatfoot | interventions — Durapatite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Osteotomy (Experimental): Using hydroxyapatite bone graft material
  Interventions: Procedure: Hydroxyapatite

INTERVENTIONS:
Procedure: Hydroxyapatite — Use of artifical bonegraft material

SUMMARY:
In this foot deformity (plano valgus) surgery may be indicated. The deformity is corrected with an osteotomy at the heelbone. In most cases bone graft material has to be obtained from the iliac crest to support the osteotomy. In the planned study a group of children will be operated with an artificial bone graft material and thus avoiding the need harvesting of bone graft at the iliac crest.

DETAILED DESCRIPTION:
Planovalgus or flatfoot deformity is observed in children with different neuromuscular disorders and is associated with pain and gait disorders due to non-reducible talonavicular joint subluxation. Surgical treatment is aimed at correcting foot malalignement and achieving sufficient plantar flexion in the ankle joint. With a calcaneal lengthening osteotomy procedure the planovalgus deformity can be corrected but it requires the use of graft material to be inserted as a bone wedge at the osteotomy site. In this way the talonavicular joint is indirectly reduced. Obtaining autograft material from the iliac crest in growing children carries a risk of growth arrest and iliac wing deformity which has led to widespread use of allograft bone when performing the operation.

New materials are being developed as substitutes for bone graft material with biphasic calcium phosphate ceramic (BCP) being the most commonly used. BCP is a mixture of porous hydroxyapatite (HA) and β-tricalcium phosphate (β -TCP). Calcium phosphate ceramics have excellent biocompatibility and are thought to be able to facilitate and guide new bone growth. This has been demonstrated in experimental studies. In retrospective clinical studies on patients having filled large bone defects with hydroxyapatite graft material radiological healing is seen at follow ups after average 7.9 years. It has also previously been demonstrated that BCP can be used as artificial bone graft in osteotomies with a good result and complete healing of the osteotomi.

ELIGIBILITY:
Inclusion Criteria:

* Flatfoot condition needing surgery

Exclusion Criteria:

* Traumatic conditions

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Healing of osteotomy | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Martin Gottliebsen, PhD-student, Principal Investigator — Aarhus University Hospital